CLINICAL TRIAL: NCT02523560
Title: Applying Telemedicine Technologies in a Novel Model of Organizing and Implementing Comprehensive Cardiac Rehabilitation in Heart Failure Patients - TELEREH-HF
Brief Title: Applying Telemedicine in a Model of Implementing Cardiac Rehabilitation in Heart Failure Patients
Acronym: TELEREH-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Collaborators: National Center for Research and Development, Poland (Other)
Responsible Party: Principal Investigator, Dr Ewa Piotrowicz, MD, PhD, National Institute of Cardiology, Warsaw, Poland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STRATEGME1/233547/13/NCBR/2015
Record Dates: First submitted 2015-08-03; First posted 2015-08-14 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Chronic Heart Failure
Keywords: Telerehabilitation; Home Monitoring; Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- telerehabilitation group (Experimental): 1 week hospital rehabilitation and 8 weeks home-based telerehabilitation and telemanagement (including HomeMonitoring)
  Interventions: Other: home-based telerehabilitation
- control group (No Intervention): Patients qualified to the control group will undergo a 9-week procedure appropriate to their clinical condition/status standardized for a particular center (usual care).

INTERVENTIONS:
Other: home-based telerehabilitation — Patients qualified to the study group will undergo, at five medical units a 9-week program of early hybrid, comprehensive cardiac telerehabilitation.
  Arms: telerehabilitation group

SUMMARY:
Applying modern technology of data collecting, monitoring, transmitting and analyzing in order to implement a novel (hybrid) model of comprehensive home-based cardiac rehabilitation in heart failure patients.

DETAILED DESCRIPTION:
Heart failure (HF) epidemic is an aggressively developing phenomenon, stimulated by developing civilization and generating worrying economic and social effects. Early comprehensive cardiac rehabilitation (CCR) is an accepted method of preventing and treating adverse cardiac events, which allows for care cost reduction. In Poland, CCR availability is highly unsatisfactory (around 8%) and unacceptably varied (0.5-70%). With the existing organization and technical background, improving this situation seems impossible. Project objective: To apply telemedicine technologies to implement a novel model of home-based CCR in HF patients.

The program, performed in six centers, will comprise 850 HF patients (randomization 1:1), in NYHA class I-III, EF≤40%, clinically stable, after a hospitalization incident. The study group patients will undergo a 9-week rehabilitation program consisting of two stages: Stage I - preliminary (one week at stationary ward), Stage II - main (8 weeks of home-based telerehabilitation). The primary end-point (days alive and out of hospital) will be assessed during a 24-month follow-up in both groups. The project will enable early secondary prevention in the population of people with HF to be implemented. It will be achieved via:

* Novel concept - "From Hospital To Home"
* Novel technology - telemedicine
* Novel method of CCR implementation

ELIGIBILITY:
Inclusion Criteria:

* patients of either sex with any aetiology of left ventricular systolic HF [as defined in the European Society of Cardiology (ESC) guidelines]
* with a left ventricular ejection fraction (LVEF) ≤40% on echocardiography;
* in New York Heart Association (NYHA) class I, II or III;
* who are to have had a hospitalization incident, be stable clinically (a patient does not need intravenous medication or has not had therapy modified for at least 7 days);
* who has no contraindications to undergo cardiopulmonary exercise test and
* who are able to exercise using the new model of home-based telerehabilitation.

Exclusion Criteria:

* NYHA class IV;
* unstable angina;
* unstable clinical status
* a history of acute coronary syndrome within the last forty days in patients with LVEF ≤35%; percutaneous angioplasty (PCI) within the last 2 weeks, coronary artery bypass grafting within the last 3 months, or initiation of cardiac resynchronization therapy (CRT-P, CRT-D) and/or implantable cardioverter-defibrillator (ICD) or pacemaker within the last six weeks;
* lack of ICD, CRT-P or CRT-D therapy despite the indications for implantation according to ESC guidelines;
* intracardiac thrombus
* rest heart rate (HR) >90/min,
* tachypnoea >20 breaths per minute
* symptomatic and/or exercise-induced cardiac arrhythmia or conduction disturbances;
* acute myocarditis and/or pericarditis
* valvular or congenital heart disease requiring surgical treatment;
* hypertrophic cardiomyopathy;
* severe pulmonary disease;
* uncontrolled hypertension;
* anemia (haemoglobin <11.0 g/dL);
* physical disability related to severe musculoskeletal or neurological problems;
* recent embolism;
* thrombophlebitis;
* acute or chronic inflammatory disease;
* acute or chronic decompensated non-cardiac diseases (thyreotoxicosis, uncontrolled diabetes)
* active malignant neoplastic diseases with survival prognosis below 2 - 5 years;
* orthotropic heart transplant in anamnesis;
* aortic aneurysm;
* severe psychiatric disorder; and
* patient's refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
days alive and out of hospital | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Piotrowicz, MD, Study Director — Institute of Cardiology, Telecardiology Center, Warsaw, Poland; Grzegorz Opolski, Prof, Study Chair — Warsaw Medical University, Department of Cardiology, Poland
Locations (5):
- Poland (5):
  - Gdański Uniwersytet Medyczny, Gdansk
  - Klinika Chorób Wewnętrznych i Rehabilitacji Kardiologicznej, Lodz
  - Warsaw Medical University; Department of Cardiology, Warsaw
  - Institute of Cardiology, Warsaw
  - Slaskie Centrum Chorób Serca, Zabrze

REFERENCES:
- [Derived] Mierzynska A, Jaworska I, Piotrowicz R, Kowalik I, Pencina M, Opolski G, Zareba W, Banach M, Orzechowski P, Glowczynska R, Szalewska D, Pluta S, Kalarus Z, Irzmanski R, Piotrowicz E. The Influence of Hybrid Comprehensive Telerehabilitation on Anxiety in Heart Failure Patients: The TELEREH-HF Randomized Clinical Trial. J Clin Psychol Med Settings. 2024 Jun;31(2):403-416. doi: 10.1007/s10880-023-09985-x. Epub 2023 Dec 18. PMID 38108961
- [Derived] Yang Z, Jia X, Li J, Mei Z, Yang L, Yan C, Han Y. Efficacy and Safety of Hybrid Comprehensive Telerehabilitation (HCTR) for Cardiac Rehabilitation in Patients with Cardiovascular Disease: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Occup Ther Int. 2023 Aug 9;2023:5147805. doi: 10.1155/2023/5147805. eCollection 2023. PMID 37593110
- [Derived] Glowczynska R, Piotrowicz E, Szalewska D, Piotrowicz R, Kowalik I, Pencina MJ, Zareba W, Banach M, Orzechowski P, Pluta S, Irzmanski R, Kalarus Z, Opolski G. Effects of hybrid comprehensive telerehabilitation on cardiopulmonary capacity in heart failure patients depending on diabetes mellitus: subanalysis of the TELEREH-HF randomized clinical trial. Cardiovasc Diabetol. 2021 May 13;20(1):106. doi: 10.1186/s12933-021-01292-9. PMID 33985509
- [Derived] Piotrowicz E, Pencina MJ, Opolski G, Zareba W, Banach M, Kowalik I, Orzechowski P, Szalewska D, Pluta S, Glowczynska R, Irzmanski R, Oreziak A, Kalarus Z, Lewicka E, Cacko A, Mierzynska A, Piotrowicz R. Effects of a 9-Week Hybrid Comprehensive Telerehabilitation Program on Long-term Outcomes in Patients With Heart Failure: The Telerehabilitation in Heart Failure Patients (TELEREH-HF) Randomized Clinical Trial. JAMA Cardiol. 2020 Mar 1;5(3):300-308. doi: 10.1001/jamacardio.2019.5006. PMID 31734701
- [Derived] Piotrowicz E, Piotrowicz R, Opolski G, Pencina M, Banach M, Zareba W. Hybrid comprehensive telerehabilitation in heart failure patients (TELEREH-HF): A randomized, multicenter, prospective, open-label, parallel group controlled trial-Study design and description of the intervention. Am Heart J. 2019 Nov;217:148-158. doi: 10.1016/j.ahj.2019.08.015. Epub 2019 Aug 22. PMID 31654944